CLINICAL TRIAL: NCT04737213
Title: An Open-label, Exploratory Study Assessing the Feasibility of SGM-101, a Fluorochrome-labeled Anti-carcinoembryonic Antigen Monoclonal Antibody for the Intraoperative Detection of Lung Metastasis in Colorectal Cancer
Brief Title: SGM-101 in Colorectal Lung Metastases
Acronym: SGM-CLM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Surgimab (Industry)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P19.101
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer; Metastatic Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective inclusion patients with colorectal lung metastases. Al injected with SGM-101.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SGM-101 (Experimental): Patients included with colorectal lung metastases, SGM-101 7.5-12.5mg, 3-5 days prior to surgery
  Interventions: Drug: SGM-101

INTERVENTIONS:
Drug: SGM-101 — Fluorescence guided surgery

SUMMARY:
Near-infrared fluorescence-guided oncologic surgery (FGOS) with the use of a tumor specific tracer (SGM-101) developed by Surgimab can provide valuable intra-operative information about tumor location and extensiveness. SGM-101 already proven to be safe and valuable in colorectal cancer.

This study aims to prove feasibility for colorectal lung metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure;
2. Patients aged over 18 years old;
3. All women of child bearing potential and all males must practice effective contraception during the study and be willing and able to continue contraception for at least 30 days after their last dose of study treatment.
4. Has the ability to communicate well with the Investigator in the Dutch language and willing to comply with the study restrictions.
5. Diagnosed with lung metastasis of colorectal origin and scheduled for a resection.

Exclusion Criteria:

1. History of any anaphylactic reaction;
2. Other malignancies either currently active or diagnosed in the last 5 years, except adequately treated in situ carcinoma of the cervix and basal or squamous cell skin carcinoma;
3. Laboratory abnormalities defined as:

   1. Aspartate AminoTransferase, Alanine AminoTransferase, Gamma Glutamyl Transferase) or Alkaline Phosphatase levels above 5 times the or;
   2. Total bilirubin above 2 times the ULN or;
   3. Serum creatinine above 1.5 times the ULN or;
   4. Platelet count below 100 x 109/L or;
   5. Hemoglobin below 4 mmol/L (females) or below 5 mmol/l (males);
   6. Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody or patients with untreated serious infections;
4. Patients pregnant or breastfeeding (pregnancy should be ruled out by a pregnancy test within two weeks prior to administration of the conjugate);
5. Any condition that the investigator considers to be potentially jeopardizing the patient's well-being or the study objectives.
6. Previous SGM-101 use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Ability of SGM-101 and a near-infrared camera system to detect colorectal lung metastases. | peroperative
  Intraoperative imaging of colorectal lung metastases based on the tumor-to-background ratio

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meijer RPJ, Galema HA, Faber RA, Bijlstra OD, Maat APWM, Cailler F, Braun J, Keereweer S, Hilling DE, Burggraaf J, Vahrmeijer AL, Hutteman M; SGM-CLM study group. Intraoperative molecular imaging of colorectal lung metastases with SGM-101: a feasibility study. Eur J Nucl Med Mol Imaging. 2024 Aug;51(10):2970-2979. doi: 10.1007/s00259-023-06365-3. Epub 2023 Aug 8. PMID 37552367